CLINICAL TRIAL: NCT03843372
Title: High Flow Nasal Cannula Compared to Continuous Positive Airway Pressure in the Treatment of Obstructive Sleep Apnea
Brief Title: High Flow Nasal Cannula for Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung-Chieh, Yu (Other)
Responsible Party: Sponsor-Investigator, Chung-Chieh, Yu, Director of Sleep Center, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201601844B0
Record Dates: First submitted 2019-02-09; First posted 2019-02-18 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Continuous Positive Airway pressure; High Flow Nasal Cannula
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: All of participants will be randomly allocated into two groups as random number table. The first group will ongoing CPAP therapy in first night and high flow nasal cannula in the second night. The second group will oppositely performed high flow nasal cannula in first night and CPAP in second night.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First night HFNC group (Experimental): The first night will receive high flow nasal cannula (HFNC) therapy and the second night accept continuous positive airway pressure (CPAP) therapy.
  Interventions: Device: High flow nasal cannula
- First night CPAP group (Active Comparator): In contrast, the first night will receive continuous positive airway pressure and the second accept high flow nasal cannula therapy.
  Interventions: Device: High flow nasal cannula

INTERVENTIONS:
Device: High flow nasal cannula — All of participants will be received one night high flow nasal cannula and another night for continuous positive airway pressure.
  Other Names: continuous positive airway pressure

SUMMARY:
This study compare the efficacy of high flow nasal cannula with nasal continuous positive airway pressure. All of participants will be randomized to receive one night high flow nasal cannula therapy and another night for nasal continuous positive airway pressure.

DETAILED DESCRIPTION:
Obstructive sleep apnea-hypopnea syndrome (OSAHS) is a common medical condition. Nasal continuous positive airway pressure (CPAP) is mainstay of treatment for OSAHS, but CPAP has some limitations. Patient who has bulbar dysfunction and poor consciousness are contraindications for CPAP. They are also not suitable for other therapy. There are still large number of patients could not accept CPAP. Alternative treatment method transnasal high flow was developed and previous study showed moderately reduce respiratory event. It is deliver 20 L/minute constant room air by nasal cannula. Because the technical limitation, the maximal flow rate is also 20 L/minute and it limit the effectiveness.

Recently, new high flow nasal cannula(HFNC) is developed. This HFNC has already widely been used for respiratory disease. It can deliver air flow up to 60 L/mins. It is also can maintain high humidifier and adequate temperature. The every 10 L/min air flow could generate approximately 1 cmH2O positive end expiratory pressure (PEEP). The higher air flow could generate more high PEEP and may have better effect than previous HFNC, but there are no study to evaluate the efficacy in OSAHS patient. Thus, the purpose of our study is to compare the efficacy of HFNC with standard CPAP therapy.

All of the participants were randomized into two groups for minimized first night effects. All of them would receive one-night HFNC therapy and another night for CPAP titration under PSG monitoring. The duration between these two treatments was approximately one week apart. The first group underwent CPAP titration on the first night and HFNC titration on the second night. Conversely, the second group was subjected to HFNC on the first night and CPAP titration on the second night. All of the participants were asked and recorded their side effects following completion of an HFNC or CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Apnea hypopnea index greater than 5 times per hour
* Age greater than 18 years old.

Exclusion Criteria:

* Central sleep apnea
* Hypoventilation syndrome
* Chronic obstructive airway disease
* Receive soft palate surgery or used an oral appliance
* Intolerance to transnasal high flow or CPAP
* Pregnant women
* Unstable hemodynamic state
* Eastern Cooperative Oncology Group Performance Status higher than grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sleep center, Principal Investigator — Chang Gung Memorial Hospital, Keelung
Locations (1):
- Sleep center, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified participants raw data will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will available within 12 months of study completion
Access Criteria: Requestors need application and explain the purpose. The data access will be provided after approved by review panel.

REFERENCES:
- [Derived] Yu CC, Huang CY, Hua CC, Wu HP. High-flow nasal cannula compared with continuous positive airway pressure in the treatment of obstructive sleep apnea. Sleep Breath. 2022 Jun;26(2):549-558. doi: 10.1007/s11325-021-02413-0. Epub 2021 Jun 18. PMID 34145538

RESULTS

PARTICIPANT FLOW:
Groups:
- HFNC First, Then CPAP: Participants first received high flow nasal cannula (HFNC) for one night. After a washout period of one week, they then received continuous positive airway pressure (CPAP) for one night.
- CPAP First, Then HFNC: Participants first received continuous positive airway pressure (CPAP) for one night. After a washout period of one week, they then received high flow nasal cannula (HFNC) for one night.
Period: Overall Study
Arm/Group | HFNC First, Then CPAP | CPAP First, Then HFNC
Started | 14 | 18
Completed | 12 | 16
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- First Night CPAP Group: The first night will receive continuous positive airway pressure(CPAP) and the second accept high flow nasal cannula(HFNC) therapy.
- Total: Total of all reporting groups
Arm/Group | First Night HFNC Group | First Night CPAP Group | Total
Number analyzed (Participants) | 12 | 16 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53.5 [43.75 to 60.75] | 53.5 [40.5 to 62] | 53.5 [42.25 to 60.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 16 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 12 | 16 | 28
BMI [Median (Inter-Quartile Range); unit: kg/m^2] — BMI(body mass index)
  kg/m^2 | 30.1 [25.47 to 34.2] | 26.95 [23.03 to 27.63] | 27.4 [24.1 to 30.8]
Neck circumference [Median (Inter-Quartile Range); unit: cm] | 41.5 [36.88 to 45] | 37.5 [35.63 to 40.75] | 38.5 [36.13 to 42.38]
AHI [Median (Inter-Quartile Range); unit: events per hour] — Apnea hypopnea index (AHI) was represented by the number of apnea and hypopnea events per hour of sleep. An apnea is defined as a drop in the peak signal excursion by 90% of the pre-event baseline, and the duration of the 90% drop in sensor signal is 10 seconds. Events are considered hypopneas when the peak signal excursions drop by 30% of the pre-event baseline, and the duration of the 30% drop in signal excursion occurs for at least 10 seconds. Hypopneas are generally associated with a 3% oxygen desaturation or cause electroencephalogram arousal.
  events per hour | 51.65 [19.23 to 65.38] | 26.9 [17.48 to 50.55] | 34.9 [18.68 to 56.13]
DI [Median (Inter-Quartile Range); unit: events per hour] — The desaturation index (DI) was the average number of desaturation episodes per hour. Desaturation episodes were defined as a decrease in the mean oxygen saturation of ≥3% from the pre-event baseline.
  events per hour | 45.15 [11.18 to 69.1] | 24.45 [12.33 to 49.53] | 29.4 [12 to 57.3]
Sleep efficiency [Median (Inter-Quartile Range); unit: %] — Sleep efficiency was the percentage of the total time spent asleep compared to the total amount of recording time.
  % | 80.7 [63.58 to 87.45] | 80.4 [78.18 to 83.23] | 80.4 [77.38 to 85.8]
Total sleep time [Median (Inter-Quartile Range); unit: minutes] — The total amount of sleep time spent during a study period.
  minutes | 324 [271 to 350] | 331.65 [315.53 to 346] | 330.15 [301.3 to 346.75]

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index
Description: The Apnea Hypopnea Index(AHI) is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. The AHI under one night transnasal high flow therapy will be compared with one night continuous positive airway pressure.
Time Frame: 2 days
Measure: Median (Inter-Quartile Range); unit: events per hour
Groups:
- CPAP: The polysomnography data of 28 participants treated with one night CPAP.
- HFNC: The polysomnography data of 28 participants received one night HFNC therapy.
Arm/Group | CPAP | HFNC
Number analyzed (Participants) | 28 | 28
events per hour | 6.15 [2.63 to 8.28] | 14.85 [6.85 to 27.3]
Statistical Analysis 1: Comparison: CPAP vs HFNC; The AHI was not a normal distribution. In the event that no carry over effect was detected between interventions, a Wilcoxon rank sum test was to be used to compare AHI between CPAP and HFNC; Test type: Superiority; p < 0.001, Wilcoxon rank sum test

2. Primary Outcome: Oxygen Desaturation Index
Description: The oxygen desaturation index (ODI) is the number of times per hour of sleep that the blood's oxygen level drop by 3% degree from baseline.The ODI under one night transnasal high flow therapy will be compared with one night continuous positive airway pressure.
Time Frame: 2 days
Measure: Median (Inter-Quartile Range); unit: events per hour
Arm/Group | CPAP | HFNC
Number analyzed (Participants) | 28 | 28
events per hour | 1.25 [0.4 to 4] | 5.25 [2.08 to 21.55]
Statistical Analysis 1: Comparison: CPAP vs HFNC; The oxygen desaturation index was not a normal distribution. In the event that no carry over effect was detected between interventions, a Wilcoxon rank sum test was to be used to compare oxygen desaturation index between CPAP and HFNC; Test type: Superiority; p < 0.001, Wilcoxon rank sum test

3. Secondary Outcome: Total Sleep Time
Description: The total amount of sleep time spent during a study period.
Time Frame: 2 days
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | CPAP | HFNC
Number analyzed (Participants) | 28 | 28
minutes | 343 [333.25 to 366.5] | 292.75 [265.63 to 325]
Statistical Analysis 1: Comparison: CPAP vs HFNC; The total sleep time was not a normal distribution. In the event that no carry over effect was detected between interventions, a Wilcoxon rank sum test was to be used to compare total sleep time between CPAP and HFNC; Test type: Superiority; p < 0.001, Wilcoxon rank sum test

4. Secondary Outcome: Sleep Efficiency
Description: Sleep efficiency is the percentage of the total time spent asleep compared to the total amount of recording time.
Time Frame: 2days
Measure: Median (Inter-Quartile Range); unit: percentage of sleep time
Arm/Group | CPAP | HFNC
Number analyzed (Participants) | 28 | 28
percentage of sleep time | 86.1 [80.15 to 90.43] | 74.25 [65.8 to 80.75]
Statistical Analysis 1: Comparison: CPAP vs HFNC; The sleep efficiency was not a normal distribution. In the event that no carry over effect was detected between interventions, a Wilcoxon rank sum test was to be used to compare sleep efficiency between CPAP and HFNC; Test type: Superiority; p = 0.008, Wilcoxon rank sum test

ADVERSE EVENTS:
Time Frame: 2 days; All of the participants were asked and recorded their side effects following completion of an HFNC or CPAP.
Description: CPAP and HFNC have been widely used in clinical practice for long time, but the serious adverse effects or mortality events are rarely reported . Our study excluded the participants who have unstable clinical condition. Therefore, there was no serious adverse events or mortality in our study.
Groups:
- CPAP: The polysomnography data of 28 participants received one night CPAP therapy.
Arm/Group | CPAP | HFNC
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 10/28 | 24/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CPAP (N=28) | HFNC (N=28)
Too strong airflow (Product Issues) | 0 | 5
CPAP Mask or HFNC cannula discomfort (Product Issues) | 6 | 1
Frequent awakenings (General disorders) | 2 | 5
Too hot airflow (Product Issues) | 0 | 5
Nasal stuffiness (General disorders) | 0 | 6
dry nose or throat (General disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03843372/Prot_SAP_000.pdf